CLINICAL TRIAL: NCT00353600
Title: Delaying the Progression of Diabetic Nephropathy in Pima Indians
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999994034; OH94-DK-N034
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-08-16

CONDITIONS: Diabetic Nephropathy
Keywords: Proteinuria; Renal Failure; Angiotension Converting Enzyme Inhibitor; Glomerular Filtration Rate
MeSH Terms: conditions — Diabetic Nephropathies; Proteinuria; Renal Insufficiency

SUMMARY:
A clinical intervention will be performed in adult diabetic Pima Indians with proteinuria to determine if an angiotensin converting enzyme (ACE) inhibitor is effective in slowing the progression of renal disease in persons with overt diabetic nephropathy attributable to type 2 diabetes mellitus (NIDDM).

The study will be conducted in the Gila River Indian Community and include proteinuric subjects selected from the Diabetic Renal Disease Study (DRDS; NIH Protocol Number 88-DK-79) in whom glomerular function has been measured at six-monthly intervals for the past 48 months. Twenty-five subjects (12 men, 13 women) aged 31-64 years are eligible for this study. These subjects all have urinary albumin-to-creatinine rations >=300 mg/g (equivalent to 300 mg albumin/day), serum creatinine concentrations < 3.0 mg/dl, and no evidence of nondiabetic renal diseases. Their GFR slopes average -0.49 ml/min/month (95% confidence interval, -0.91 to -0.07), and 11 of them (8 men, 3 women) are hypertensive (systolic blood pressure >=140 mm Hg, diastolic blood pressure >=90 mm Hg).

Subjects will be treated with an ACE inhibitor, and measurements of glomerular filtration rate (GFR) and renal plasma flow (RPF) will be made at six monthly intervals until the subjects' progress to renal failure. GFR slope (ml.min/month) will be computed, and the slope prior to the initiation of an ACE inhibitor will be compared with that obtained during treatment.

DETAILED DESCRIPTION:
A clinical intervention will be performed in adult diabetic Pima Indians with proteinuria to determine if an angiotensin converting enzyme (ACE) inhibitor is effective in slowing the progression of renal disease in persons with overt diabetic nephropathy attributable to type 2 diabetes mellitus.

The study will be conducted in the Gila River Indian Community and include proteinuric subjects selected from the Diabetic Renal Disease Study (DRDS; NIH Protocol Number 88-DK-79) in whom glomerular function has been measured at six-monthly intervals for the past 48 months. Twenty-five subjects (12 men, 13 women) aged 31-64 years are eligible for this study. These subjects all have urinary albumin-to-creatinine ratios greater than or equal to 300 mg/g (equivalent to 300 mg albumin/day), serum creatinine concentrations less than 3.0 mg/dl, and no evidence of nondiabetic renal diseases. Their GFR slopes average -0.49 ml/min/month (95 percent confidence interval, -0.91 to -0.07), and 11 of them (8 men, 3 women) are hypertensive (systolic blood pressure greater than or equal to 140 mm Hg, diastolic blood pressure greater than or equal to 90 mm Hg).

Subjects will be treated with an ACE inhibitor, and measurements of glomerular filtration rate (GFR) and renal plasma flow (RPF) will be made at six monthly intervals until the subjects' progress to renal failure. GFR slope (ml/min/month) will be computed, and the slope prior to the initiation of an ACE inhibitor will be compared with that obtained during treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for participation in the study, subjects must meet the following criteria:

Previous completion of the DRDS;

Serum creatinine concentration less than 3.0 mg/dl;

Serum potassium concentration less than or equal to 5.7 mEq/L;

At least 2 of 3 screening urinary albumin-to-creatinine ratios greater than or equal to 300 mg/g;

Willingness, after receiving a thorough explanation of the study, to participate.

Severe hypertension will not affect eligibility for the study.

EXCLUSION CRITERIA:

In addition to the criteria outlined in the DRDS protocol, subjects with the following characteristics will be excluded:

Pregnancy. Women of childbearing age and not surgically sterilized must have a negative pregnancy test prior to entry and prior to each renal clearance study.

Hypersensitivity to ACE inhibitors.

Conditions that are likely to interfere with informed consent or compliance with the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1994-08-19; Study Completion 2011-08-16

CONTACTS AND LOCATIONS:
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Background] Anderson S, Rennke HG, Garcia DL, Brenner BM. Short and long term effects of antihypertensive therapy in the diabetic rat. Kidney Int. 1989 Oct;36(4):526-36. doi: 10.1038/ki.1989.227. PMID 2681929
- [Background] Zatz R, Dunn BR, Meyer TW, Anderson S, Rennke HG, Brenner BM. Prevention of diabetic glomerulopathy by pharmacological amelioration of glomerular capillary hypertension. J Clin Invest. 1986 Jun;77(6):1925-30. doi: 10.1172/JCI112521. PMID 3011862
- [Background] Zatz R, Meyer TW, Rennke HG, Brenner BM. Predominance of hemodynamic rather than metabolic factors in the pathogenesis of diabetic glomerulopathy. Proc Natl Acad Sci U S A. 1985 Sep;82(17):5963-7. doi: 10.1073/pnas.82.17.5963. PMID 3862110